CLINICAL TRIAL: NCT05867251
Title: A Phase 1/2, First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of AVZO-021 as a Single Agent and in Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: Study of AVZO-021 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avenzo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVZO-021-1001
Record Dates: First submitted 2023-04-13; First posted 2023-05-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor; HR+/HER2- Breast Cancer; HR+, HER2-, Advanced Breast Cancer; CCNE1 Amplification; Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Endometrial Cancer; TNBC - Triple-Negative Breast Cancer
Keywords: Advanced solid tumor; HR+/HER2- Breast Cancer; Breast Cancer; Advanced Breast Cancer; CCNE1 Amplification; Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Endometrial Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Endometrial Neoplasms; Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — palbociclib; Fulvestrant; Letrozole; ribociclib; abemaciclib; Carboplatin; sacituzumab govitecan

STUDY DESIGN:
Intervention Model Description: Phase 1 dose-escalation Phase 2 dose-expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1, monotherapy (Part 1A) (Experimental): Escalating doses of once daily, oral AVZO-021 in 28-day cycles.
  Interventions: Drug: AVZO-021
- Phase 1, combination (Parts 1B and 1C) (Experimental): Escalating doses of once daily, oral AVZO-021 in 28-day cycles starting at least 1 DL below the monotherapy MTD/RP2D dose in combination with:
  1B1) fulvestrant
  1B2) palbociclib plus either fulvestrant or letrozole
  1B3) ribociclib plus either fulvestrant or letrozole
  1B4) abemaciclib plus either fulvestrant or letrozole
  1B5) sacituzumab govitecan-hziy
  1C) carboplatin
  Interventions: Drug: AVZO-021; Drug: Palbociclib; Drug: Fulvestrant; Drug: Letrozole; Drug: Ribociclib; Drug: Abemaciclib; Drug: Carboplatin; Drug: Sacituzumab Govitecan-hziy
- Phase 2, monotherapy (Part 2A) (Experimental): Oral doses of AVZO-021 in 28-day cycles at the RP2D determined in Part 1A.
  Interventions: Drug: AVZO-021
- Phase 2, combination (Parts 2B and 2C) (Experimental): Oral doses of AVZO-021 in 28-day cycles at the RP2D determined in Parts 1B/1C, in combination with:
  2B1) fulvestrant
  2B2) palbociclib plus either fulvestrant or letrozole
  2B3) ribociclib plus either fulvestrant or letrozole
  2B4) abemaciclib plus either fulvestrant or letrozole
  2B5) sacituzumab govitecan-hziy
  2C) carboplatin
  Interventions: Drug: AVZO-021; Drug: Palbociclib; Drug: Fulvestrant; Drug: Letrozole; Drug: Ribociclib; Drug: Abemaciclib; Drug: Carboplatin; Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: AVZO-021 — AVZO-021 is a selective and potent oral inhibitor of CDK2 being developed for the treatment of patients with advanced solid tumors with CDK2 dependency (1A), CCNE1 amplified solid tumors (2A), HR+/HER2- BC (1B1-1B5, 2B1-2B5) and CCNE1 amplified EOC (1C, 2C)
Drug: Palbociclib — Antineoplastic agent, cyclin-dependent kinase 4/6 inhibitor
  Other Names: Ibrance
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)
Drug: Fulvestrant — Antineoplastic agent, estrogen receptor antagonist
  Other Names: Faslodex
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)
Drug: Letrozole — Antineoplastic agent, aromatase inhibitor
  Other Names: Femara
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)
Drug: Ribociclib — Antineoplastic CDK4/6 inhibitor
  Other Names: Kisqali
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)
Drug: Abemaciclib — Antineoplastic CDK4/6 inhibitor
  Other Names: Verzenio
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)
Drug: Carboplatin — Alkylating agent
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)
Drug: Sacituzumab Govitecan-hziy — Trop-2 antibody and topoisomerase inhibitor
  Other Names: Trodelvy
  Arms: Phase 1, combination (Parts 1B and 1C); Phase 2, combination (Parts 2B and 2C)

SUMMARY:
This study, the first clinical trial of AVZO-021, aims to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, maximum tolerated dose, and anti-tumor effects of AVZO-021 in patients with advanced solid tumors. AVZO-021 is an oral medication that inhibits cyclin-dependent kinase 2 (CDK 2).

DETAILED DESCRIPTION:
AVZO-021 is a compound being developed for the treatment of patients with advanced solid tumors, specifically, HR+/HER2- breast cancer and cyclin E1 (CCNE1) altered malignancies. AVZO-021 is a selective and potent cyclin-dependent kinase 2 (CDK2) inhibitor, which plays an important role in cell cycle regulation. This is a Phase 1/2 first-in-human, open-label, nonrandomized, multicenter study of AVZO-021. Phase 1 is a dose-escalation phase aimed at assessing the safety and tolerability of AVZO-021 and determining the recommended phase 2 dose (RP2D) as monotherapy and combination therapy. Phase 2 is a dose-expansion phase that will be conducted to assess the antitumor activity of AVZO-021 as monotherapy and combination therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged ≥18 years old at screening with Eastern Cooperative Oncology Group (ECOG) 0-1.
2. Disease-related inclusion criteria by study phase and part:

   i) Phase 1a Monotherapy Dose Escalation: Patients with locally advanced or metastatic HR+/HER2- breast cancer, CCNE1-amplified tumors that are either epithelial ovarian cancer, primary peritoneal cancer, fallopian tube cancer, endometrial cancer or TNBC, with no other oncogenic driver mutations that are treatable and standard therapies are no longer effective, appropriate, or safe in the opinion of the investigator and medical monitor. Patients with any additional tumor type with CCNE1 amplification can be enrolled only if clinical data is supportive and approved by medical monitor (Cohort 1A).

   ii) Phase 1b Combination Dose Escalation: histologically or cytologically confirmed diagnosis of locally advanced or metastatic HR+ HER2- (HER2-low may be allowed if failed standard of care therapy) breast cancer, who have been previously treated with inhibitor of CDK4/6 and endocrine therapy(Cohorts 1B1, 1B2, 1B3, 1B4, and 1B5); or histologically or cytologically confirmed diagnosis of CCNE1- amplified, locally advanced or metastatic, platinum-refractory or platinum-resistant EOC, primary peritoneal, or fallopian tube cancer (Cohort 1C).

   iii) Phase 2a Monotherapy dose expansion: Histologically or cytologically confirmed diagnosis of locally advanced or metastatic CCNE1 amplified epithelial ovarian cancer, primary peritoneal cancer, fallopian tube cancer, endometrial cancer or TNBC, with no other oncogenic driver mutations that are treatable and standard therapies are no longer effective, appropriate, or safe in the opinion of the investigator and medical monitor (Cohort 2A).

   iv) Phase 2b Combination dose expansion: Histologically or cytologically confirmed diagnosis of locally advanced or metastatic HR+/HER2- (HER2-low may be allowed if failed standard of care therapy) breast cancer who have been previously treated with no more than 1 prior CDK4/6 inhibitor and endocrine therapy (Cohorts 2B1, 2B2, 2B3, 2B4, and 2B5); or Histologically or cytologically confirmed diagnosis of locally advanced or metastatic, CCNE1-amplified, platinum-refractory or platinum-resistant EOC, primary peritoneal cancer, or fallopian tube cancer (Cohort 2C).
3. No more than 2 prior cytotoxic chemotherapy regimens for locally advanced/metastatic disease (excepting patients treated with an antibody-drug conjugate, with ovarian cancer if there disease is platinum resistant or refractory, having progressed beyond all SOC care; and patients who have received prior chemotherapy in the adjuvant or neoadjuvant setting >12 months prior to starting AVZO-021 treatment).
4. Measurable disease as determined by RECIST version 1.1.
5. Adequate bone marrow and organ function.
6. Ability to swallow capsules or tablets.

Key Exclusion Criteria:

1. Received an investigational agent or anticancer therapy within 2 weeks, or 5 half-lives of the drug, whichever is shorter, prior to planned start of AVZO-021.
2. Received any CDK2 inhibitor, protein kinase membrane associated tyrosine/threonine 1 (PKMYT1) inhibitor, or WEE1 inhibitor anticancer therapy. For cohort B5, prior therapy with topoisomerase inhibitors is not permitted.
3. Undergone major surgery within 4 weeks prior to planned start of AVZO-021.
4. Received radiotherapy for palliation within 7 days of the first dose of study treatment, unless specified otherwise in the protocol.
5. Active CNS metastases or confirmed leptomeningeal disease are not eligible.
6. Unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade >1 at the time of starting study treatment.
7. Clinically unstable cardiac function as described in the protocol.
8. Any active or chronic infection/disease that compromises the immune system.
9. Current treatment with strong or moderate cytochrome P450 (CYP)3A4 inhibitors or inducers.
10. Active second malignancy unless in remission with life expectancy > 2 years and with documented sponsor approval.
11. Pregnancy, lactation, or plans to breastfeed during the study or within 6 months of the last dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLTs) during the first cycle (Phase 1) | 28 Days
  Number of participants with DLTs assessed for severity using CTCAE v5.0 criteria will be summarized by dose level.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and lab abnormalities (Phase 1) | Approximately 22 months
  To evaluate the type, incidence, severity, timing, seriousness, and relationship to study treatment of adverse events and any laboratory abnormalities summarized by dose level.
Determination of Recommended Phase 2 Dose (RP2D) (Phase 1) | Approximately 16 months
  RP2D for AVZO-021 is less than or the same as the maximum tolerated dose (MTD) as defined by the occurrence of DLTs and TEAEs calculated using isotonic regression.
Objective Response Rate (ORR) (Phase 2) | Approximately 52 months
  Defined as the proportion of patients with a confirmed Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Progression Free Survival (PFS) (Phase 2) | Approximately 52 months
  Defined as the time from study drug treatment to death or disease progression, as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Overall Survival (OS) (Phase 2) | Approximately 76 months
  Defined as the time from study drug treatment initiation to death from any cause.
Duration of response (DOR) (Phase 2) | Approximately 52 months
  Defined as the time from the first confirmed response to radiologic/objective progression.

SECONDARY OUTCOMES:
PK Parameters: Maximum plasma concentration (Cmax) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Time to maximum plasma concentration (Tmax) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Area under the plasma concentration-time curve from time 0 to last measurable concentration (AUC 0-last) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Area under the plasma concentration-time curve from time 0 to last measurable concentration (AUC 0-tau) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Minimum observed plasma concentration at steady state (Cmin, ss) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Accumulation ration (Rac) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Elimination half-life (t1/2) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Apparent clearance (CL/F) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
PK Parameters: Apparent volume of distribution during terminal phase (Vz/F) (monotherapy and combination) | Cycle 1 days 1, 2, 8, 14, and 15 (each cycle is 28 days)
Evaluate the effect of a high-fat meal on the PK of AVZO-021 (Phase 1) | 5 days

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - Providence Cancer Institute, Portland, Oregon
  - Sidney Kimmel Cancer Center (SKCC) at Jefferson Health, Philadelphia, Pennsylvania
  - Texas Oncology - DFW, Dallas, Texas
  - NEXT Virginia, Fairfax, Virginia
- Australia (2):
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales

IPD SHARING:
Plan to Share IPD: No